CLINICAL TRIAL: NCT02056236
Title: TELSTAR: Treatment of ELectroencephalographic STatus Epilepticus After Cardiopulmonary Resuscitation
Acronym: TELSTAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Twente (Other)
Collaborators: Rijnstate Hospital (Other); Medisch Spectrum Twente (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Radboud University Medical Center (Other); University Medical Center Groningen (Other); St. Antonius Hospital (Other); VieCuri Medical Centre (Other); Université Libre de Bruxelles (Other); Maasstad Hospital (Other); Maastricht University Medical Center (Other); Canisius-Wilhelmina Hospital (Other)
Responsible Party: Principal Investigator, Jeannette Hofmeijer, MD PhD, University of Twente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEF-14-18; NL46296.044.13 (Other: VCMO the Netherlands)
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Arrest; Anoxic Encephalopathy; Status Epilepticus
Keywords: Cardiac arrest; Postanoxic encephalopathy; Electroencephalographic status epilepticus; EEG monitoring; Anti-epileptic drugs
MeSH Terms: conditions — Heart Arrest; Hypoxia, Brain; Status Epilepticus | interventions — Lorazepam; Midazolam; Propofol; Levetiracetam; Valproic Acid; Thiopental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anti-epileptic drugs (Experimental): Step 1: Phenytoin (loading dose 15-20 mg/kg iv, maintenance doses 150 mg iv twice per day) PLUS one of the following benzodiazepines (bolus + continuous infusion): lorazepam or midazolam. Benzodiazepine dosing regimes should be based on national and local protocols for status epilepticus treatment
  Step 2: Propofol infusion (with a maximum rate of 8 mg/kg/hour) PLUS a second anti-epileptic drug in addition to fenytoin: Option 1: levetiracetam bolus 1500 mg, followed by 1000 mg 2 dd 1 intravenously or Option 2: valproic acid bolus 10-20 mg/kg in 30 min, followed by15 mg/kg/day in 2 dosages intravenously.
  Step 3: Thiopental, initial dosage 12,5 mg/kg/hr for the first 6 hours followed by 5 mg/kg/hr for 6 hours. After these loading dosages, treatment should be guided by the EEG pattern.
  Interventions: Drug: Anti-epileptic drugs
- No anti-epileptic drugs (Active Comparator): The non-intervention group will be treated conform standard guidelines of treatment of comatose patients after cardiac arrest, but without anti-epileptic drugs or EEG based deep sedation. Treatment to suppress clinical myoclonia or seizures with low dose propofol is left to the discretion of the treating physician.
  Decisions regarding limitation or withdrawal of treatment will be done in accordance with the Dutch guideline "postanoxic coma" in both treatment arms. Reasons for withdrawal of treatment will be documented.
  Interventions: Other: No anti-epileptic drugs

INTERVENTIONS:
Drug: Anti-epileptic drugs — Recommendations for the treatment of status epilepticus are based on recent international guidelines for treatment of overt status epilepticus.
  The objective of treatment with AED is to suppress all epileptiform activity. There is no clear proof that induction of a burst-suppression pattern is of additional value and induction of burst suppression is therefore not obligate. If the electroencephalographic status epilepticus returns after tapering sedative treatment at 24 hours, the procedure will be repeated. If the status returns after 2 x 24 hours, it will be considered refractory.
  Decisions regarding limitation or withdrawal of treatment will be done in accordance with the Dutch guideline "postanoxic coma". Reasons for withdrawal of treatment will be documented.
  Other Names: Lorazepam; Midazolam; Fenytoin; Propofol; Levetiracetam; Valproate; Thiopental
  Arms: Anti-epileptic drugs
Other: No anti-epileptic drugs — The non-intervention group will be treated conform standard guidelines of treatment of comatose patients after cardiac arrest, but without anti-epileptic drugs or EEG based deep sedation. Treatment to suppress clinical myoclonia or seizures with low dose propofol is left to the discretion of the treating physician.
  Decisions regarding limitation or withdrawal of treatment will be done in accordance with the Dutch guideline "postanoxic coma". Reasons for withdrawal of treatment will be documented.
  Arms: No anti-epileptic drugs

SUMMARY:
The purpose of this study is to estimate the effect of medical treatment of electro-encephalographic status epilepticus on neurological outcome of patients with postanoxic encephalopathy after cardiac arrest.

DETAILED DESCRIPTION:
Rationale: Electroencephalographic status epilepticus is described in 9-35% of patients with postanoxic encephalopathy after cardiac arrest and is associated with case fatality rates of 90-100%. It is unclear whether (some) electroencephalographic seizure patterns in these patients represent a condition which can be treated with antiepileptic drugs to improve outcome, or have to be regarded as an expression of severe ischemic damage, in which treatment with antiepileptic would be futile. Therefore, both treatment with and treatment without antiepileptic drugs are considered standard modalities in these patients. We aim to compare these standard strategies and hypothesize that aggressive and early treatment of electro-encephalographic status epilepticus with antiepileptic drugs improves outcome as compared to treatment without these drugs.

Objective: To estimate the effect of medical treatment of electro-encephalographic status epilepticus on neurological outcome of patients with postanoxic encephalopathy after cardiac arrest

Study design: We will perform a multicenter clinical trial with randomized treatment allocation, open label treatment and blinded endpoint evaluation (PROBE design). The intervention contrast will be aggressive medical treatment vs. no treatment of electroencephalographic status epilepticus, in addition to standard best medical management of comatose patients after cardiac arrest, including mild therapeutic hypothermia.

Study population: The study population will consist of adult patients with postanoxic encephalopathy after cardiac arrest, admitted to the intensive care unit, with electroencephalographic status epilepticus on continuous EEG, who are eligile for inclusion in this trial.

Intervention: Treatment of electroencephalographic status epilepticus will be based on guidelines for treatment of overt status epilepticus. The objective of this treatment will be to suppress all epileptiform activity in the EEG. If the electroencephalographic status epilepticus will return after tapering sedative treatment at 24 hours, the procedure will be repeated. If the status will return after 2 x 24 hours, it will be considered refractory.

Main study parameters/endpoints: The primary outcome measure will be neurological outcome defined as the score on the Cerebral Performance Category (CPC) at 3 months dichotomized as good (CPC 1-2 = no or moderate neurological disability) and poor (CPC 3-5 = severe disability, coma, or death).

Sample size: With a presumed reduction of poor outcome of 7%, from 99% - 92%, alpha of 5%, power of 80%, one tailed testing, and one interim analysis by an independent data safety and monitoring board, the objected number of inclusions is 172. With an estimation of an incidence of electroencephalographic status epilepticus of 20% in patients with postanoxic coma, the total number of patients to be monitored will be 860.

Nature and extent of the burden and risks associated with participation: Medical treatment of electroencephalographic status epilepticus may modify the high risk of death. Otherwise, this treatment of electroencephalographic status epilepticus may lead to prolonged hospitalization of several days of comatose patients that otherwise would have died. The risk of an increase of morbidity or mortality on the longer term is considered negligible.

ELIGIBILITY:
Inclusion Criteria:

* Patients after cardiac arrest with suspected postanoxic encephalopathy
* Age 18 years or older
* Continuous EEG with at least eight electrodes started within 24 hours after cardiac arrest
* Electroencephalographic status epilepticus on continuous EEG
* Possibility to start treatment within three hours after detection of electroencephalographic status epilepticus.

Exclusion Criteria:

* A known history of another medical condition with limited life expectancy (<6 months)
* Any progressive brain illness, such as a brain tumor or neurodegenerative disease
* Pre-admission Glasgow Outcome Scale score of 3 or lower
* Reason other than neurological condition to withdraw treatment
* Follow-up impossible due to logistic reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2014-04; Primary Completion 2021-04-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Neurological outcome | three months
  The primary outcome measure will be neurological outcome defined as the score on the Cerebral Performance Category (CPC) at 3 months dichotomized as good (CPC 1-2 = no or moderate neurological disability) and poor (CPC 3-5 = severe disability, coma, or death).

SECONDARY OUTCOMES:
Long term outcome | 12 months
  Secondary outcome measures will include i) mortality; ii) the CPC score at 6 and 12 months; iii) length of stay on the ICU; iv) duration of mechanical ventilation; v) seizure recurrence within one year; vi) quality of life as measured by the Medical Outcomes Study 36-item short-form health survey (SF36), depression as measured by the Montgomery and Åsberg Depression Rating Scale (MADRS) , and cognitive functioning as measured by detailed neuropsychological examination after 12 months.
  Secondary outcome measures in survivors will be collected to thoroughly assess outcome and quality of life of survivors. These outcome measures will not be collected to test between-group differences, since the estimated number of survivors is small.
  Furthermore, a limited amount of data on the use of resources will be collected for analysis of cost-effectiveness, including place of residence at one year and admission in hospitals, rehabilitations centers, and nursing homes within the first year.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette Hofmeijer, MD PhD, Principal Investigator — Rijnstate Hospital and University of Twente; Michel van Putten, MD PhD, Principal Investigator — Medisch Spectrum Twente and University of Twente; Janneke Horn, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Barry Ruijter, MD, Study Director — University of Twente
Locations (11):
- Hôpital Erasme - Université libre de Bruxelles, Brussels, Lenniksebaan 808, Belgium
- Netherlands (10):
  - Radboud University Medical Center, Nijmegen, Geert Grooteplein-Zuid 10
  - Medisch Spectrum Twente, Enschede, Haaksbergerstraat 55
  - University Medical Center Groningen, Groningen, Hanzeplein 1
  - St. Antonius Hospital, Nieuwegein, Koekoekslaan 1
  - Academic Medical Center, Amsterdam, Meibergdreef 9
  - Maasstad Hospital, Rotterdam, South Holland
  - VieCuri Medical Centre, Venlo, Tegelseweg 210
  - Rijnstate Hospital, Arnhem, Wagnerlaan 55
  - Maastricht UMC+, Maastricht
  - Canisius-Wilhelmina Hospital, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruijter BJ, van Putten MJ, Horn J, Blans MJ, Beishuizen A, van Rootselaar AF, Hofmeijer J; TELSTAR study group. Treatment of electroencephalographic status epilepticus after cardiopulmonary resuscitation (TELSTAR): study protocol for a randomized controlled trial. Trials. 2014 Nov 6;15:433. doi: 10.1186/1745-6215-15-433. PMID 25377067
- [Derived] van Putten MJAM, Ruijter BJ, Horn J, van Rootselaar AF, Tromp SC, van Kranen-Mastenbroek V, Gaspard N, Hofmeijer J; TELSTAR Investigators. Quantitative Characterization of Rhythmic and Periodic EEG Patterns in Patients in a Coma After Cardiac Arrest and Association With Outcome. Neurology. 2024 Aug 13;103(3):e209608. doi: 10.1212/WNL.0000000000209608. Epub 2024 Jul 11. PMID 38991197
- [Derived] Ruijter BJ, Keijzer HM, Tjepkema-Cloostermans MC, Blans MJ, Beishuizen A, Tromp SC, Scholten E, Horn J, van Rootselaar AF, Admiraal MM, van den Bergh WM, Elting JJ, Foudraine NA, Kornips FHM, van Kranen-Mastenbroek VHJM, Rouhl RPW, Thomeer EC, Moudrous W, Nijhuis FAP, Booij SJ, Hoedemaekers CWE, Doorduin J, Taccone FS, van der Palen J, van Putten MJAM, Hofmeijer J; TELSTAR Investigators. Treating Rhythmic and Periodic EEG Patterns in Comatose Survivors of Cardiac Arrest. N Engl J Med. 2022 Feb 24;386(8):724-734. doi: 10.1056/NEJMoa2115998. PMID 35196426
- [Derived] Hofmeijer J, van Putten MJ. EEG in postanoxic coma: Prognostic and diagnostic value. Clin Neurophysiol. 2016 Apr;127(4):2047-55. doi: 10.1016/j.clinph.2016.02.002. Epub 2016 Feb 11. PMID 26971488
- [Derived] Ruijter BJ, van Putten MJ, Hofmeijer J. Generalized epileptiform discharges in postanoxic encephalopathy: Quantitative characterization in relation to outcome. Epilepsia. 2015 Nov;56(11):1845-54. doi: 10.1111/epi.13202. Epub 2015 Sep 19. PMID 26384469